CLINICAL TRIAL: NCT00912223
Title: A Phase II Trial of Non-Myeloablative Allogeneic Hematopoietic Cell Transplantation for Patients With Relapsed Follicular Non-Hodgkin's Lymphoma Beyond First Complete Response (BMT CTN #0701)
Brief Title: Blood Stem Cell Transplant With Low Dose Chemotherapy for Relapsed Follicular Non-Hodgkin's Lymphoma (BMT CTN 0701)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0701; U01HL069294 (NIH); U01HL06929406 (Other: National Cancer Institute (NCI)); 5U24CA076518 (NIH); NCT00867074 (obsolete NCT alias)
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Follicular Non-Hodgkin's Lymphoma; Hematopoietic Stem Cell Transplant (HSCT); Non-Myeloablative Transplant (NST)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hematopoietic Stem Cell Transplant (Experimental): Participants will undergo a non-myeloablative allogeneic hematopoietic stem cell transplant.
  Interventions: Biological: Hematopoietic Stem Cell Transplant

INTERVENTIONS:
Biological: Hematopoietic Stem Cell Transplant — NOTE: The - sign is the number of days before the transplant and the + sign is the number of days after the transplant.
  The conditioning regimen will consist of the following:
  * Rituxan 375 mg/m^2 on Day -13
  * Rituxan 1000 mg/m^2 on Days -6, +1, and +8
  * Fludarabine 30 mg/m^2 on Days -5 to -3
  * Cyclophosphamide 750 mg/m^2 on Days -5, -4, -3
  Day 0 will be the day of the transplant.
  The GVHD prophylaxis will consist of the following:
  * Tacrolimus .09 mg/kg/po (Day -2 thru Day +180). Doses will be adjusted to maintain blood levels of 5-15 ng/mL.
  * Methotrexate 5 mg/m^2 (Days +1, +3, and +6). Unrelated donor recipients will receive a fourth dose on Day +11.

SUMMARY:
Blood stem cell transplants are one treatment option for people with lymphoma or other types of blood cancers. For this type of treatment, family members or unrelated donors with a similar tissue type usually donate their blood stem cells to the transplant patients. This study will evaluate the effectiveness of a type of blood stem cell transplant that uses lower doses of chemotherapy in people with relapsed follicular non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
Follicular NHL, a type of blood cancer, is the second most common type of non-Hodgkin's lymphoma, with approximately 15,000 new cases being diagnosed each year in the United States. Chemotherapy is a common treatment option for people with NHL, and at first most people achieve cancer remission with initial chemotherapy. However, after the initial chemotherapy, people with this disease typically experience a continuous pattern of relapse that results in progressively shorter remission durations. A blood stem cell transplant is another treatment option for people with follicular NHL. In a blood stem cell transplant procedure, healthy blood stem cells are taken from a donor and transplanted into the patient. The cells can be donated by a family member or an unrelated donor who has a similar tissue type. Typically, people who are undergoing a blood stem cell transplant receive high doses of chemotherapy before the transplant to prepare their bodies to accept the donor stem cells. In this study, participants will undergo a type of stem cell transplant called a nonmyeloablative transplant, which involves a reduced intensity method of transplantation that does not require high doses of chemotherapy. The purpose of the study is to examine the effectiveness of a nonmyeloablative allogeneic blood stem cell transplant at improving survival rates in people with relapsed follicular NHL.

This study will enroll people with relapsed follicular NHL. At a baseline study visit, participants will undergo a medical history review, physical examination, blood collection, lung function testing, computed tomography (CT) scans, a bone marrow biopsy, and questionnaires to assess quality of life. Participants will be admitted to the hospital and on various days in the 2 weeks before the transplant, they will receive fludarabine, cyclophosphamide, rituximab, which are cancer medications, and tacrolimus, a medication that will help prevent graft-versus-host disease (GVHD), which is an attack by the donor cells on the body's normal tissues. Participants will then undergo the blood stem cell transplant. At various times during the 2 weeks after the transplant, participants will receive rituximab and methotrexate, which is another medication to prevent GVHD. They will also receive tacrolimus for at least 6 months to help prevent GVHD. Participants will remain in the hospital for as long as necessary to recover from the transplant. Follow-up study visits will occur weekly for Weeks 1 to 14, and then at Months 6, 12, 18, and 24. At each study visit, select baseline procedures will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Must have confirmed CD20+ follicle center lymphoma that meets one of the following:

  1. Histologically confirmed recurrent Revised European American Lymphoma (REAL) Classification CD20+ follicle center lymphoma, follicular grades I and II
  2. Histologically confirmed World Health Organization (WHO) classification CD20+ follicular lymphoma grades 1, 2, or 3a.

     For either classification, the diffuse component of large cleaved cells (if present) cannot be greater than 50% of cellularity. Patients do not have to express t(14;18) to be eligible.
* Any number of prior regimens (including autologous hematopoietic cell transplantation [HCT]); the most recent prior regimen must have occurred more than 28 days before study entry
* Must demonstrate chemosensitive or radiosensitive disease to most recent prior regimen and meet one of the following criteria:

  1. Patients in second or subsequent complete remission (CR)
  2. Patients in first or subsequent partial remission (PR)
  3. Patients experiencing a relapse that demonstrates a response, as defined as largest nodal mass less than or equal to 3 cm or greater than or equal to 50% reduction in estimated lymph node volume measured as a product of bi-dimensional measurements (see protocol for detailed definition).
  4. Patients with stable follicular lymphoma are eligible if all lymph node masses are less than or equal to 3 cm and are smaller or unchanged in size to the most recent salvage regimen.
* Patients with human leukocyte antigen (HLA)-matched donors that meet the following criteria:

  1. 6/6 HLA-matched related donor. HLA typing must be performed by DNA methods for HLA-A and B at intermediate (or higher) resolution, and DRB1 at high resolution. The donor must be willing to donate peripheral blood stem cells and meet institutional criteria for stem cell donation. The donor must be medically eligible to donate stem cells according to individual transplant center criteria; or,
  2. 8/8 HLA-matched unrelated donor. HLA typing must be performed by DNA methods for HLA-A, B, C, and DRB1 at high resolution. The donor must be willing to donate peripheral blood stem cells and meet National Marrow Donor Program (NMDP) criteria for stem cell donation. The donor must be medically eligible to donate stem cells according to NMDP criteria.
* Patients with adequate organ function, as measured by the following:

  1. Heart: Left ventricular ejection fraction at rest greater than 45%
  2. Lungs: Diffusing capacity of the lung for carbon monoxide (DLCO), forced expiratory volume in one second (FEV1), or forced vital capacity (FVC) greater than 50% of predicted (corrected for hemoglobin). For patients in whom pulse oximetry is performed, baseline O2 saturation greater than 85% (when lung function testing cannot be performed due to age restrictions)
  3. Liver: Bilirubin less than two times the upper limit of normal for age as per local laboratory; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than three times the upper limit of normal as per local laboratory
  4. Kidney: Calculated or measured creatinine clearance greater than or equal to 40 mL/min; if creatinine is greater than or equal to 1.5 mg/dL then 24-hour urine for measured creatinine clearance should be performed.

Exclusion Criteria:

* Patients in first CR
* Karnofsky performance score less than 70%
* Patients with follicular lymphoma that demonstrates evidence of histologic transformation. In the presence of B symptoms, rapid growth of a single dominant site, or prolonged (> 2 yrs) interval since last tissue diagnosis, investigators are encouraged to consider re-biopsy of nodes prior to enrollment.
* Uncontrolled hypertension
* Uncontrolled bacterial, viral, or fungal infection (i.e., currently taking medication and progression of clinical symptoms)
* Prior cancer, other than resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent less than 5 years will not be allowed unless approved by the medical monitor or protocol chair. Cancer treated with curative intent greater than 5 years will be allowed.
* Pregnant or breastfeeding
* Seropositive for human immunodeficiency virus (HIV)
* Fertile men or women unwilling to use contraception from the time of initiation of conditioning until 6 months post-transplant
* Prior allogeneic HSCT
* Known anaphylactic reaction to rituximab
* Seropositive for any of the following: HIV ab, hepatitis B sAg or polymerase chain reaction (PCR)+, or hepatitis C ab or PCR+

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-04; Primary Completion 2014-11 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research (CIBMTR), Medical College of Wisconsin
Locations (21):
- United States (21):
  - City of Hope National Medical Center, Duarte, California
  - University of California, San Diego (UCSD) Medical Center, La Jolla, California
  - University of California, Davis Medical Center, Sacramento, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute (DFCI)/Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI)/Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, MD Anderson Cancer Research Center, Houston, Texas
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Findings will be published in a manuscript.
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Laport GG, Wu J, Logan B, Bachanova V, Hosing C, Fenske T, Longo W, Devine SM, Nademanee A, Gersten I, Horowitz M, Lazarus HM, Riches ML; Blood and Marrow Transplant Clinical Trials Network. Reduced-Intensity Conditioning with Fludarabine, Cyclophosphamide, and High-Dose Rituximab for Allogeneic Hematopoietic Cell Transplantation for Follicular Lymphoma: A Phase Two Multicenter Trial from the Blood and Marrow Transplant Clinical Trials Network. Biol Blood Marrow Transplant. 2016 Aug;22(8):1440-1448. doi: 10.1016/j.bbmt.2016.04.014. Epub 2016 Apr 23. PMID 27118571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between April 2009 and November 2012 from 21 different transplant centers.
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplant
Started | 65
Completed | 62
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Not transplanted | 1
Not completed — Transformed disease | 1

BASELINE CHARACTERISTICS:
Population: Received transplant
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
Age, Continuous [Median (Full Range); unit: years] | 55 [29 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Karnofsky Performance Score [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning on a scale of 0 - 100; where 100 equals normal quality of life with no evidence of disease, 90 equals ability to carry on normal activity with minor signs/symptoms of disease, and 80 equals normal activity with effort and some signs/symptoms of disease.
  participants
    100 | 29
    90 | 28
    80 | 5
Comorbidity Index Score [Number; unit: participants] — Comorbidity is graded on a scale of 0 to 6 based on the adjusted risk of mortality and the sum of scores result in a single comorbidity index score for a participant. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality.
  participants
    0 | 31
    1-2 | 16
    >3 | 15
Disease Status [Number; unit: participants] — Disease status is categorized best to worst by second/subsequent complete remission (CR2), first partial remission (PR1), second partial remission (PR2). Complete remission criteria is disappearance of all evidence of disease and partial remission criteria is regression of measurable disease and no new sites.
  participants
    CR2 | 32
    PR1 | 6
    ≥ PR2 | 16
    Stable Disease | 2
    Unknown | 6
Number of Prior Chemotherapy Regimens [Number; unit: participants]
  2 | 14
  3 | 16
  4 | 12
  ≥ 5 | 20
Donor Type (HLA match) [Number; unit: participants]
  Matched Related Donor (6/6 allele) | 33
  Matched Unrelated Donor (8/8 allele) | 29
Recipient Cytomegalovirus Status [Number; unit: participants]
  Positive | 35
  Negative | 27

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Patients are considered a failure for this endpoint if they die, or if they relapse/progress or receive anti-lymphoma therapy not including planned post-transplant radiation.
Time Frame: Year 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
percentage of participants | 73 [60 to 82]

2. Secondary Outcome: Graft Failure
Description: Primary graft failure is defined as a donor peripheral blood T cell chimerism < 5% at Day +30 post-transplant. Secondary Graft Failure is defined as documented engraftment followed by loss of graft as defined by donor peripheral blood T cell chimerism < 5%.
Time Frame: Day 30
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
participants
  Primary Graft Failure | 0
  Secondary Graft Failure | 0

3. Secondary Outcome: Donor Cell Engraftment
Description: Donor engraftment is defined as > 5% donor peripheral blood T cell chimerism by Day +30 post-transplant in the setting of Absolute Neutrophil Count (ANC) recovery (ANC >500/mm^3 for 3 consecutive days).
Time Frame: Days 30 and 100
Measure: Median (Full Range); unit: percentage of donor T-cell chimerism
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
percentage of donor T-cell chimerism
  Day 30 | 94 [25 to 100]
  Day 100 | 96 [25 to 100]

4. Secondary Outcome: Time to Neutrophil Recovery
Description: Neutrophil Recovery is defined as ANC > 500/mm^3 for 3 consecutive days.
Time Frame: Day 60
Measure: Median (Full Range); unit: days
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
days | 13 [8 to 48]

5. Secondary Outcome: Acute Graft-versus-Host Disease (GVHD)
Description: The event is the incidence of grades II-IV acute GVHD from day of transplant, where grade IV is worst. The first day of acute GVHD onset at a certain grade will be used to calculate a cumulative incidence curve for that acute GVHD grade. GVHD should be monitored in accordance with BMT CTN manual of procedures guidelines. Acute GVHD grading was based on the consensus conference criteria (Przepiorka, et. al., 1994) and the Center for International Blood and Marrow Transplant Research (CIBMTR) grading criteria.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
percentage of participants | 27 [16 to 39]

6. Secondary Outcome: Chronic GVHD
Description: The event is the incidence and severity of chronic GVHD from day of transplant, a cumulative incidence curve will be computed along with a 95% confidence interval at two years post-transplant. Death prior to occurrence of chronic GVHD will be considered as a competing risk.
Time Frame: Year 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
percentage of participants | 61 [48 to 74]

7. Secondary Outcome: Overall Survival
Description: The event is death from any cause.
Time Frame: Years 2 and 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
percentage of participants
  2 years | 84 [72 to 91]
  3 years | 82 [70 to 90]

8. Secondary Outcome: Treatment-related Mortality (TRM)
Description: The event is death occurring in patients in continuous complete remission. The TRM distribution will be estimated by the Kaplan-Meier curve.
Time Frame: Year 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
percentage of participants | 16 [8 to 27]

9. Secondary Outcome: Infections
Time Frame: Year 2
Population: no data collected
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 0

10. Secondary Outcome: Quality of Life
Time Frame: Year 2
Population: No data collected
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 0

11. Secondary Outcome: Immunologic Reconstitution
Description: Quantitative immunoglobulins (IgG)
Time Frame: Year 1
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
mg/dL | 431 [79 to 1430]

12. Secondary Outcome: Incidence of Toxicities
Description: Number of participants that experiences at least one grade 3 - 5 toxicity during the first two years, where grade 5 is worst. Toxicity grades are based on the NCI CTCAE Version 3.0.
Time Frame: Year 2
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 62
participants | 50

13. Secondary Outcome: Serum Rituximab (RTX) Levels
Description: RTX concentration levels within participants
Time Frame: Baseline, Days 28 and 365
Population: Serum RTX concentrations were collected at baseline (n=57), day +28 (n=56), and day +365 (n=44) for a compliance rate of 92%, 90%, and 80% at the assigned time points.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 57
ng/mL
  Baseline | 42100 [500 to 70200]
  Day 28 | 341000 [500 to 670000]
  Day 365 | 920 [500 to 122000]

ADVERSE EVENTS:
Time Frame: 3 years post-transplant
Description: Serious Adverse Events (AE) are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event. Only unexpected grades 3-5 adverse events were required to be reported through the AE system per protocol.
Arm/Group | Hematopoietic Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 2/62
Other Adverse Events (participants affected / at risk) | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplant (N=62)
Appendicitis (Infections and infestations) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-05-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT00912223/Prot_SAP_ICF_000.pdf